CLINICAL TRIAL: NCT00689403
Title: A Phase I, Two-part, Randomised, Open, Single-centre, Crossover Study to Evaluate Different Extended-release Formulations of AZD1305 When Given as Single Oral Doses to Healthy Male Volunteers
Brief Title: Evaluate Different Extended-release (ER) Tablets/Capsules of AZD1305
Acronym: 2007-005765-38
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Helen Lunde, MD, Medical Science Director, Emerging Arrhythmia and Lipids, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D3190C00014
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: AZD1305; pharmacokinetics; Properties of different ER formulations
MeSH Terms: interventions — tert-butyl (2-(7-(2-(4-cyano-2-fluorophenoxy)ethyl)-9-oxa-3,7-diazabicyclo(3.3.1)non3-yl)ethyl)carbamate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A: 2x2 crossover (Experimental): 4 different AZD1305 ER formulations
  Interventions: Drug: AZD1305
- Part B: 3x3 crossover (Experimental): 2 different AZD1305 ER formulations and a reference formulation
  Interventions: Drug: AZD1305

INTERVENTIONS:
Drug: AZD1305 — Extended release capsules, oral single doses
  Arms: Part A: 2x2 crossover
Drug: AZD1305 — Extended release capsules, oral single doses
  Arms: Part B: 3x3 crossover

SUMMARY:
To study the properties of different tablets/capsules of AZD1305 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male between the age of 20 - 45
* Non-smoking

Exclusion Criteria:

* Potassium outside normal reference values
* ECG findings outside normal range

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables | During all dosing visits

SECONDARY OUTCOMES:
Adverse events, ECG, safety laboratory, vital signs, physical examination | During the study

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lunde, MD, Study Director — AstraZeneca R&D, Mölndal, Sweden; Daniel Bradford, MD, MA, MBBS, DCPSA, Principal Investigator — PAREXEL Clinical Pharmacology Research UnitHarrow, United Kingdom
Locations (1):
- Research Site, Harrow, United Kingdom